CLINICAL TRIAL: NCT03351829
Title: Gene Therapy of Beta Thalassemia Using a Self-inactivating Lentiviral Vector
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17008
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Beta-Thalassemia
Keywords: Beta Thalassemia; Lentiviral vector; Gene
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene-modified autologous stem cells (Experimental): Autologous stem cells transduced with lentiviral vector carrying the related gene ex vivo
  Interventions: Genetic: Gene-modified autologous stem cells

INTERVENTIONS:
Genetic: Gene-modified autologous stem cells — 1 infusion for 5x10^6~1x10^7 gene-modified cells; or more infusions depending on the circumstances

SUMMARY:
This is a Phase I/II clinical trial of gene transfer for treating Beta-thalassemia using a self-inactivating lentiviral vector to functionally correct the defective gene(s). The objectives are to evaluate the safety and efficacy of the gene transfer clinical protocol.

DETAILED DESCRIPTION:
Thalassemia is considered the most common genetic disorder worldwide. Beta-thalassemia is caused by mutations in the beta-globin gene which encodes the beta-globin protein, leading to the ineffective erythropoiesis, hemolysis and anemia. Currently, the only cure for thalassemia is bone marrow transplantation from a related, compatible donor, which has, however, the significant risk of transplant related mortality, graft versus host disease and limited source. Therefore, gene transfer, achieved by transplantation of the patient's own stem cells that have been genetically-modified with the corrected gene, could potentially cure thalassemia.

This study will use an experimental gene transfer procedure performed in a laboratory to insert the related gene into the participant's autologous stem cells using a self-inactivating lentiviral vector. The purpose of this study is to evaluate the safety and effectiveness of the gene transfer procedure and to determine the ability of the gene-corrected cells at generating new, healthy blood cells in individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Beta Thalathemia.
2. Age: ≥ 4 years.
3. Karnofsky: ≥ 80%.
4. Left ventricular ejection fraction (LVEF): > 50%; no obvious heart disease and pulmonary hypertension.
5. Pulmonary function is normal; forced expiratory volumein one second (FEV1) and vital capacity greater than 60% and DLCO > 50%.
6. Serum creatinine ≤ 2 × upper limit of normal range.
7. MRI showed no super-iron load in the heart and liver, and no severe cirrhosis.
8. Normal Coagulation.
9. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Diagnosis of active malignant disease (other than Bowen disease or cervical cancer); or has family history of cancer.
2. Myelopathy, tumor-related cytogenetic changes or other more severe blood diseases.
3. Has alcoholism experience within 6 months prior to enrollment.
4. History of epilepsy.
5. History of bone marrow transplantation.
6. Existence of an available HLA-identical related donor.
7. Pregnant or lactating females.
8. Subject infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), HTLV (HTLV antibody positive), Treponema pallidum antibody positive or TB culture positive.
9. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  Physiological parameter (measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Treatment responses | 1 year
  Blood routine indexes will be got before and after treatment. Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Quality of life | 1 year
  Quality of life will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No